CLINICAL TRIAL: NCT00000726
Title: Foscarnet Treatment of Serious CMV Retinitis Infection in Patients With Acquired Immunodeficiency Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 015; FDA 20D; 10991 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Foscarnet; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
To explore the safety and usefulness of foscarnet, an antiviral agent, in the treatment of cytomegalovirus (CMV) retinitis. Untreated CMV retinitis is a rapidly progressive, blinding disease in AIDS patients. The manner in which foscarnet breaks down in the body and the effect of increasing periodic intravenous doses are also studied. Foscarnet is active in vitro (test tube) against herpes viruses, including CMV, by inhibiting the virus DNA polymerases, enzymes necessary for virus replication, without affecting cellular DNA polymerases. Opportunistic CMV disease in AIDS is usually seen as retinitis, colitis, esophagitis, hepatitis, pancreatitis, encephalitis, or pneumonia. Ganciclovir has been used to treat AIDS patients with CMV disease but can cause severe neutropenia (very low neutrophil cell counts). Foscarnet does not suppress the production of neutrophils or other leukocytes (myelosuppression) and has shown in vitro activity against HIV.

DETAILED DESCRIPTION:
Foscarnet is active in vitro (test tube) against herpes viruses, including CMV, by inhibiting the virus DNA polymerases, enzymes necessary for virus replication, without affecting cellular DNA polymerases. Opportunistic CMV disease in AIDS is usually seen as retinitis, colitis, esophagitis, hepatitis, pancreatitis, encephalitis, or pneumonia. Ganciclovir has been used to treat AIDS patients with CMV disease but can cause severe neutropenia (very low neutrophil cell counts). Foscarnet does not suppress the production of neutrophils or other leukocytes (myelosuppression) and has shown in vitro activity against HIV.

Treatment is given for a total of 10 weeks with a 2-week induction regimen followed by randomization to daily maintenance foscarnet for 8 weeks. If induction therapy is tolerated without unexpected toxicity, patients are allowed to self-administer foscarnet at home via central venous catheter and may receive up to 11 days of induction therapy by self-administration on an outpatient basis. Foscarnet will be administered in open-label fashion so that both investigator and patient will know the dose. Within the study, there are 8 patients who upon entering the 2nd week of maintenance foscarnet therapy are treated with zidovudine (AZT).

ELIGIBILITY:
Exclusion Criteria

Concurrent Medication:

Excluded:

* Acyclovir.
* Zidovudine (AZT).
* Any potentially nephrotoxic agent, especially aminoglycosides, pentamidine, or amphotericin B.

Prior Medication:

Excluded:

* Ganciclovir.
* Foscarnet.
* Excluded within 7 days of study entry:
* Any potentially nephrotoxic agent.
* Excluded within 14 days of study entry:
* Cytomegalovirus hyperimmune globulin in therapeutic doses.
* Immunomodulators.
* Biologic response modifiers.
* Investigational agents.
* Amphotericin B maintenance for a systemic mycosis.

Known allergy to foscarnet.

Active AIDS-defining opportunistic infection other than cytomegalovirus (CMV) including systemic mycosis, pulmonary or neurologic impairment (comatose).

Patient must be diagnosed as having:

* AIDS CDC Group IV.C.
* Cytomegalovirus (CMV) retinitis as identified by its characteristic ophthalmoscopic appearance and verified by fundus photography.
* One pending culture for CMV from blood and urine prior to study entry.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53
Dates: Study Completion 1992-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobson M, Study Chair
Locations (5):
- United States (5):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - USC School of Medicine / Norris Cancer Hosp, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Mem Sloan - Kettering Cancer Ctr, New York, New York

REFERENCES:
- [Background] Jacobson MA, Polsky B, Causey D, Davis R, Tong W, O'Donnell JJ, Kuppermann BD, Heinemann MH, Feinberg J, Lizak P, et al. Pharmacodynamic relationship of pharmacokinetic parameters of maintenance doses of foscarnet and clinical outcome of cytomegalovirus retinitis. Antimicrob Agents Chemother. 1994 May;38(5):1190-3. doi: 10.1128/AAC.38.5.1190. PMID 8067763
- [Background] Aweeka F, Gambertoglio J, Mills J, Jacobson MA. Pharmacokinetics of intermittently administered intravenous foscarnet in the treatment of acquired immunodeficiency syndrome patients with serious cytomegalovirus retinitis. Antimicrob Agents Chemother. 1989 May;33(5):742-5. doi: 10.1128/AAC.33.5.742. PMID 2546491
- [Background] Jacobson MA, O'Donnell JJ, Mills J. Foscarnet treatment of cytomegalovirus retinitis in patients with the acquired immunodeficiency syndrome. Antimicrob Agents Chemother. 1989 May;33(5):736-41. doi: 10.1128/AAC.33.5.736. PMID 2546490
- [Background] Jacobson MA, Crowe S, Levy J, Aweeka F, Gambertoglio J, McManus N, Mills J. Effect of Foscarnet therapy on infection with human immunodeficiency virus in patients with AIDS. J Infect Dis. 1988 Oct;158(4):862-5. No abstract available. PMID 2844921
- [Background] Jacobson MA, Causey D, Polsky B, Hardy D, Chown M, Davis R, O'Donnell JJ, Kuppermann BD, Heinemann MH, Holland GN, et al. A dose-ranging study of daily maintenance intravenous foscarnet therapy for cytomegalovirus retinitis in AIDS. J Infect Dis. 1993 Aug;168(2):444-8. doi: 10.1093/infdis/168.2.444. PMID 8393058
- [Background] Jacobson MA, Causey D, Polsky B, Hardy D, Feinberg JE, O'Donnell JJ, Kuppermann BD, Heinemann MH, Holland G, Mills J. Dose-ranging study of daily intravenous (IV) maintenance foscarnet (PFA) therapy (Rx) for cytomegalovirus (CMV) retinitis in AIDS patients (ACTG protocol 015/915). Int Conf AIDS. 1990 Jun 20-23;6(2):113 (abstract no FB96)
- [Background] Jacobson MA, Causey D, Hardy D, Polsky B, Mills J, Feinberg JE. Tolerance and efficacy of daily intravenous (IV) maintenance foscarnet (PFA) therapy for cytomegalovirus (CMV) retinitis in AIDS patients (ACTG protocol 015). Int Conf AIDS. 1989 Jun 4-9;5:242 (abstract no MBP123)